CLINICAL TRIAL: NCT07062991
Title: Effects of Kendall Exercises Versus Scapular Stabilization Exercises on Neck Pain, Range of Motion and Neck Disability in Mechanical Neck Pain
Brief Title: Effects of Kendall Exercises Versus Scapular Stabilization Exercises Oin Mechanical Neck Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR &AHS/24/0158 Neelam
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Neck Pain
Keywords: Pain; Disability; Mobilization Technique
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kendall Exercises (Experimental): Kendall exercises which includes:
  Chin tuck in supine Stretching the cervical extensors Shoulder retraction with theraband Stretching of the pectoralis major muscle Every strengthening exercise will be repeated for 12 repetitions and done for 3 sets and each stretching exercise will be hold for 30 seconds and repeated 3 times. The exercises will be performed three times per week for 4 weeks
  Interventions: Other: Kendall Exercises
- Scapular stabilization exercises (Experimental): Scapular stabilization exercises which includes:
  Shoulder shrugs Prone arm lift Stretching of levator scapular Stretching pectoralis minor muscle Each strengthening exercise will be repeated for 15 repetitions of 3 sets and each stretching exercises will be hold for 30 seconds and repeated 3 times. The exercises will be performed three days per week for 4 weeks.
  Interventions: Other: Scapular stabilization exercises

INTERVENTIONS:
Other: Kendall Exercises — Kendall exercises which includes: Chin tuck in supine Stretching the cervical extensors Shoulder retraction with theraband Stretching of the pectoralis major muscle Every strengthening exercise will be repeated for 12 repetitions and done for 3 sets and each stretching exercise will be hold for 30 seconds and repeated 3 times. The exercises will be performed three times per week for 4 weeks
  Arms: Kendall Exercises
Other: Scapular stabilization exercises — Shoulder shrugs Prone arm lift Stretching of levator scapular Stretching pectoralis minor muscle Each strengthening exercise will be repeated for 15 repetitions of 3 sets and each stretching exercises will be hold for 30 seconds and repeated 3 times. The exercises will be performed three days per week for 4 weeks.
  Arms: Scapular stabilization exercises

SUMMARY:
Neck pain is a multifactorial disease, and is a major problem in modern society. Patients with NCNP usually have alterations in cervical proprioception and PS. They may also develop symptoms such as dizziness or vertigo. A recently published study shows that patients with NCNP suffer greater sensations of stunning and lack of proprioception than patients with benign paroxysmal vertigo.

DETAILED DESCRIPTION:
This study will be a randomized controlled trial and will be conducted on general population in Gujrat. Non-probability convenient sampling will be used to collect the data. Sample size of 48 subjects with age group between 25-45 years will be taken. Data will be collected from the patients having present complaint of Nonspecific Neck pain. Outcome measures will be taken using Numeric pain rating scale (NPRS) for pain, Neck disability index (NDI) for measuring disability and goniometer for range of motion (ROM). An informed consent will be taken. Subjects will be selected based on inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. Both the Groups will receive standard physical therapy, while Group A will receive bruegger's exercises and Group B will receive Upper thoracic mobilization. Outcome measures will be measured at baseline then after 4 weeks(post). Data analysis will be done by SPSS version 21.

ELIGIBILITY:
Inclusion Criteria:

* Male and females between 20-40 years of age, Patients having pain that had persisted for 12 weeks or more,
* Patients with generalized neck pain provoked by sustained neck postures, neck movements, pain on palpation of cervical musculature without any pathologies.

Exclusion Criteria:

* History of whiplash injury,
* Cervical surgery,
* Fracture of the cervical or scapular and Neurological impairments

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | upto 4 weeks
  The Numeric Pain Rating Scale (NPRS) is perhaps the most frequently applied scale used to quantify pain intensity in the clinical setting. It is an 11-point numeric scale, ranging from 0 indicating no pain to 10 indicating worst pain imaginable
Universal Goniometer (UG) | upto 4 weeks
  The cervical flexion, extension, side bending, and rotation range of motion will be measured through universal goniometer. The universal goniometer is frequently used to quantify limitations in ROM. Physical therapists use the ROM measurement to quantify limitations at the beginning of intervention and to quantify the effects of intervention.
Neck disability index (NDI) | upto 4 weeks
  NDI consists of 10 items: pain intensity, personal care, lifting, reading, headache, concentration, work, sleeping, driving, and recreation. Each item consists of six score levels that range from zero to five points.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nugraha MHS, Antari N, Saraswati N. The efficacy of muscle energy technique in individuals with mechanical neck pain: a systematic review. Sport Fit J. 2020;8:91-8.
- [Background] Heggannavar A, Battula L. Immediate effect of thoracic distraction thrust versus upper thoracic crossed hand manipulation in mechanical neck pain: A randomized clinical trial. Physiotherapy-The Journal of Indian Association of Physiotherapists. 2021;15(1):22-7.
- [Background] Junaid M, Yaqoob I, Shakil Ur Rehman S, Ghous M. Effects of post-isometric relaxation, myofascial trigger point release and routine physical therapy in management of acute mechanical neck pain: a randomized controlled trial. J Pak Med Assoc. 2020 Oct;70(10):1688-1692. doi: 10.5455/JPMA.15939. PMID 33159734
- [Background] Choudhary S, Hussain ME, Moscovitch A, Pandi-Perumal SR, Bahammam AS. Multimodal physiotherapy improves pain, functional disability, sleep quality and health related quality of life in chronic mechanical neck pain patients. International Journal of Health Science Research. 2021;8(3):138-48.
- [Background] Ganu S, Gor U. Effects of abdominal control feedback and scapular stabilization exercise on chronic neck pain. International Journal of Health Sciences and Research. 2021;11(6):318-25.
- [Background] Ashfaq M, Babur MN, Malick WH, Hussain MA, Awan WA. Comparative effectiveness of proprioceptive neuromuscular facilitation and passive vertebral mobilization for neck disability in patients with mechanical neck pain: A randomized controlled trial. J Bodyw Mov Ther. 2022 Jul;31:16-21. doi: 10.1016/j.jbmt.2022.02.009. Epub 2022 Mar 18. PMID 35710215
- [Background] Seo YG, Park WH, Lee CS, Kang KC, Min KB, Lee SM, Yoo JC. Is Scapular Stabilization Exercise Effective for Managing Nonspecific Chronic Neck Pain?: A Systematic Review. Asian Spine J. 2020 Feb;14(1):122-129. doi: 10.31616/asj.2019.0055. Epub 2019 Nov 1. PMID 31668049